CLINICAL TRIAL: NCT07140068
Title: Comparing GumChucks Flossing System and Interdental Brushes in Plaque Removal Efficacy Among Lebanese Adolescents (A Randomized Controlled Trial).
Brief Title: GumChucks vs Interdental Brushes in Plaque Removal.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Principal Investigator, Rim Daher, Principal Investigator, Pediatric Dentistry Resident, Beirut Arab University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-H-0120-D-M-0527
Record Dates: First submitted 2025-08-16; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Adolescent; Dental Plaque; Gingivitis; Oral Hygiene; Pediatric Dentistry
Keywords: Dental plaque; Gingivitis; Oral hygiene; Flossing; Interdental brushes; Interdental cleaning; Dental floss; Oral health; Preventive dentistry; Adolescents
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial using a split-mouth design, where each participant's mouth was divided into two halves, one side assigned to the GumChucks flossing system and the other side to interdental brushes.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded to which side of each participant's mouth received the handled flossing system or interdental brush. Participants and care providers were not masked due to the visible nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GumChucks Flossing System (Experimental): Participants cleaned all interdental spaces on one side of the mouth using the handled flossing system (GumChucks®) twice daily after toothbrushing with a medium- bristle toothbrush and fluoride toothpaste. The proper C-shape flossing technique was demonstrated, and written instructions were provided.
  Interventions: Device: Handled dental flossing system (GumChucks®)
- Interdental Brush (Experimental): Participants cleaned all interdental spaces on the other side of the mouth using appropriately sized interdental brushes twice daily after toothbrushing with a medium-bristle toothbrush and fluoride toothpaste. Proper technique was demonstrated, and written instructions were provided.
  Interventions: Device: Interdental Brush

INTERVENTIONS:
Device: Handled dental flossing system (GumChucks®) — Handled dental flossing system (GumChucks®) designed for easier C-shape flossing. Participants were instructed to clean all interdental spaces on the assigned side twice daily after toothbrushing with fluoride toothpaste using a medium-bristle toothbrush. Proper technique was demonstrated and written instructions provided.
  Arms: GumChucks Flossing System
Device: Interdental Brush — Appropriately sized interdental brushes for cleaning interdental spaces on the assigned side. Participants were instructed to clean twice daily after toothbrushing with fluoride toothpaste using a medium-bristle toothbrush. Proper technique was demonstrated and written instructions provided.
  Arms: Interdental Brush

SUMMARY:
This study compared two ways of cleaning between the teeth, Gumchucks (a new handled dental flossing system) and interdental brushes, in Lebanese adolescents aged 10-15 years.

Plaque is a soft layer of bacteria that can build up between teeth and cause tooth decay and gum problems. Toothbrushing alone cannot always clean these spaces. Extra cleaning tools, such as floss or interdental brushes, are recommended. Gumchucks uses two small handles to hold the floss, making it easier to use, especially for children. It had not previously been directly compared with interdental brushes in this age group.

In this study, 60 healthy adolescents were included to use Gumchucks on one side of their mouth and interdental brushes on the other side for six months. They were asked to clean twice daily after toothbrushing.

Researchers measured plaque levels between teeth, gum bleeding, time taken to clean, and which method participants and parents preferred The goal was to find out which method worked better and was preferred, to help dentists recommend the best way for young people to keep their teeth and gums healthy.

DETAILED DESCRIPTION:
This randomized, parallel, split-mouth, examiner-blind clinical trial compared Gumchucks, a handled dental flossing system, and interdental brushes in removing interdental plaque and reducing gingival inflammation in Lebanese adolescents.

Participants were 60 healthy adolescents aged 10-15 years, each with at least four posterior interdental contacts and no recent antibiotic or antibacterial mouth rinse use. In each participant, one side of the mouth was randomly assigned to Gumchucks and the other side to interdental brushing. Participants cleaned twice daily after brushing with fluoride toothpaste using a medium toothbrush.

During the first session, dental prophylaxis was performed, the correct size of interdental brush was selected for each participant, and demonstrations and written instructions for both devices were provided. The cleaning time was measured in seconds for each participant using each device, and the preferences were collected from participants and parents using 5-point Likert scale questionnaires at the end of the first session. Participants were then asked to avoid interdental cleaning for three days before the baseline assessment.

Clinical assessments performed at baseline, 1 month, 3 months, and 6 months included the Papillary Bleeding Index (PBI) (scored 0-4 at mesio-facial, disto-facial, mesio-lingual/palatal, and disto-lingual/palatal sites of interdental papillae) and the Quigley Hein Plaque Index (modified by Turesky): scored 0-5 at the same sites after using a plaque disclosing agent.

Intra- and inter-examiner reliability were evaluated using Cohen's Kappa statistics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents (ASA 1) aged between 10 and 15 years;
* Patients who had at least 4 posterior interdental contacts;
* Patients who were able to follow verbal and/or written instructions, where they were asked to perform what they understood directly after reading the written instructions and listening to the explanation.

Exclusion Criteria:

* Patients who had antibiotics within the last 6 months;
* Patients who were using antibacterial mouth rinses;
* Patients with physical, intellectual, developmental, or emotional disabilities;
* Patients with unilateral mastication or a nonfunctional side.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Interdental plaque removal | Baseline, 1 month, 3 months, and 6 months.
  Evaluated by measuring the modified Quigley-Hein plaque index scores (by Turesky et al., 1970) after using a plaque disclosing agent.
Gingival inflammation reduction | Baseline, 1 month, 3 months, and 6 months.
  Evaluated by measuring the papillary bleeding index (PBI) scores (by Mühlemann, 1977).

SECONDARY OUTCOMES:
Cleaning time | Dental Prophylaxis Session, 3 days before the Baseline examination session
  Measured during the Dental Prophylaxis Session, after receiving the dental prophylaxis and the instructions on C-shape flossing with GumChucks and proper use of interdental brushes. The principal investigator recorded the total time for each participant to clean all interdental contacts on the phone's stopwatch in seconds, using both products each at a time, in front of a mirror.
Participant and Parent Preferences. | Dental Prophylaxis Session, 3 days before the Baseline examination session
  Preferences toward the use of GumChucks in comparison to interdental brush were measured by a 5-point Likert scale questionnaire at the end of the Dental Prophylaxis Session, after using both products and measuring the cleaning time. The answers ranged between strongly disagree and strongly agree. The adolescent participants' questionnaire asked if GumChucks helped to clean interdentally faster and more frequently and if it was easier to use and more preferred over interdental brush. The parents' questionnaire asked if GumChucks was easier for their children as well as for them to help their children clean interdentally, if their children would clean interdentally more often, and if they would buy GumChucks for their children.

CONTACTS AND LOCATIONS:
Overall Officials: Rim K Daher, Masters, Principal Investigator — Beirut Arab University
Locations (1):
- Beirut Arab University, Beirut, Tarik El Jadida, Lebanon

IPD SHARING:
Plan to Share IPD: No
This study will only share aggregate results, such as mean plaque scores, cleaning times, and preference percentages, in publications. Individual participant-level data (IPD) will not be shared.